CLINICAL TRIAL: NCT03296007
Title: Evaluating the Psychophysiological Effects of a Smartphone-Based Mindfulness Task on Individuals With Clinically Significant Symptoms of Chronic Pain, Depression and Anxiety
Brief Title: Evaluating the Psychophysiological Effects of a Smartphone-Based Mindfulness Task
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: York University (Other)
Responsible Party: Principal Investigator, Joel Katz, Professor, York University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: #e2017 - 303
Record Dates: First submitted 2017-09-22; First posted 2017-09-28 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Chronic Pain; Depression, Anxiety
MeSH Terms: conditions — Chronic Pain; Depression; Anxiety Disorders | interventions — Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Meditation App (Experimental): Participants randomized to this arm will use a smartphone app to practice mindfulness meditation for 12 minutes.
  Interventions: Behavioral: Mindfulness Meditation
- Mindfulness Meditation No App (Active Comparator): Participants randomized to this arm will not use a smartphone app, but will receive instructions to practice mindfulness meditation for 12 minutes.
  Interventions: Behavioral: Mindfulness Meditation

INTERVENTIONS:
Behavioral: Mindfulness Meditation — A meditative practice involving paying attention to present moment experiences and focusing on breathing sensations.

SUMMARY:
The aim of the present study is to evaluate the psychophysiological effects of a smart phone based mindfulness meditation app (MMA) for individuals with clinically significant symptoms of major depression and/or anxiety, or symptoms of chronic pain. Specifically, the study aims to examine parasympathetic tone using HRV (primary outcome), mind-wandering and present awareness, mood symptoms, and breath focus in groups of participants who self-report clinically significant symptoms of depression and/or anxiety (DA), chronic pain symptoms (CP), as well as control participants who do not meet our criteria for either (Controls (C). All study groups will be randomized to a mindfulness meditation app (MMA+) condition or a mindfulness meditation condition without the app (MMA-) after a brief stress-induction procedure.

ELIGIBILITY:
Inclusion Criteria:

* York University students

Exclusion Criteria:

* Individuals with diagnosed cardiac conditions (e.g. coronary artery disease, arrhythmias etc) will be excluded due to confounds with heart rate variability assessment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2016 (Actual)
Dates: Start 2017-11-10 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Heart Rate Variability | 22 minutes
  A stress biomarker derived from heart rate recordings that reflects parasympathetic control of cardiac output

CONTACTS AND LOCATIONS:
Overall Officials: Joel Katz, PhD, Principal Investigator — York University
Locations (1):
- York University, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Azam MA, Latman VV, Katz J. Effects of a 12-Minute Smartphone-Based Mindful Breathing Task on Heart Rate Variability for Students With Clinically Relevant Chronic Pain, Depression, and Anxiety: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2019 Dec 2;8(12):e14119. doi: 10.2196/14119. PMID 31789601